CLINICAL TRIAL: NCT07244419
Title: Emapalumab for the Prevention of Graft Rejection in Hematopoietic Stem Cell Transplant (HSCT) Recipients
Brief Title: Prevention of Graft Rejection in Hematopoietic Stem Cell Transplant (HSCT) Recipients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Sobi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-0167
Record Dates: First submitted 2024-10-30; First posted 2025-11-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic Stem Cell Transplantation; Graft Failure
MeSH Terms: interventions — Emapalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Emapalumab 3 mg/kg (Active Comparator): Patients randomized to this arm will receive 3mg/kg of emapalumab intravenously (IV) once on day +1 after HSCT. Up to two additional, 10mg/kg rescue doses may be administered if patients developed signs and symptoms of acute graft rejection. Rescue dose administration decisions will be made in consultation with the lead study investigator. Emapalumab is a ligand-based therapy, which means high levels of circulating ligand (i.e. interferon gamma) will rapidly consume the drug. For these reasons, rescue doses may be given as early as 24 hours from the prior dose.
  Interventions: Drug: Emapalumab 3 mg/kg
- Emapalumab 10 mg/kg (Active Comparator): Patients randomized to this arm will receive 10mg/kg of emapalumab intravenously (IV) once on day +1 after HSCT. Up to two additional, 10mg/kg rescue doses may be administered if patients developed signs and symptoms of acute graft rejection. Rescue dose administration decisions will be made in consultation with the lead study investigator. Emapalumab is a ligand-based therapy, which means high levels of circulating ligand (i.e. interferon gamma) will rapidly consume the drug. For these reasons, rescue doses may be given as early as 24 hours from the prior dose.
  Interventions: Drug: Emapalumab 10 mg/kg

INTERVENTIONS:
Drug: Emapalumab 3 mg/kg — Subjects will be randomized to either receive a 3mg/kg or 10mg/kg intravenous dose of emapalumab once and may receive up to two additional doses if clinical concern for impending graft rejection develops.
  Arms: Emapalumab 3 mg/kg
Drug: Emapalumab 10 mg/kg — Subjects will be randomized to either receive a 3mg/kg or 10mg/kg intravenous dose of emapalumab once and may receive up to two additional doses if clinical concern for impending graft rejection develops.
  Arms: Emapalumab 10 mg/kg

SUMMARY:
The investigators hypothesize that graft rejection after hematopoietic stem cell transplant (HSCT) is primarily driven by interferon gamma, and prophylactic interferon gamma inhibition in high-risk patients will prevent graft rejection. Additionally, knowledge of emapalumab PK/PD and in vitro mechanistic effects of emapalumab in this novel setting will guide optimization of dosing regimens and treatment approaches in future studies.

DETAILED DESCRIPTION:
Graft rejection is a devastating and understudied complication of hematopoietic stem cell transplant (HSCT) due to the lack of available interventions outside of re-transplantation. Re-transplantation is challenging and is associated with increased morbidity and mortality.

The purpose of this study is to learn more about emapalumab and its ability to prevent graft rejection in hematopoietic stem cell transplant (HSCT) recipients. Specifically, the study doctors would like to learn more about the efficacy and treatment of emapalumab as a prophylactic intervention for graft rejection.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing allogeneic HSCT at our institution will be evaluated for graft rejection risk factors. Patients deemed high risk for graft rejection will have 2 or more of the following: mismatched or haploidentical donor, ex vivo t-cell depleted graft, prior history of graft rejection.

Exclusion Criteria:

* Known hypersensitivity to any constituent of the study medication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Preliminary efficacy of Emapalumab | 100 days
  Measured by the incidence of graft rejection in the treatment cohort.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of emapalumab after 10 mg/kg prophylactic dosing | Until day 42 or time of rescue dose, whichever is sooner
  * Measured by the Cmax (ng/mL) of emapalumab after 10mg/kg dose
  * Cmax values will be calculated using every 48 hour blood collections beginning at the time of emapalumab administration (day 1 after HSCT) until day 21.
Maximum plasma concentration of emapalumab after 3 mg/kg prophylactic dosing | Until day 42 or time of rescue dose, whichever is sooner
  * Measured by the Cmax (ng/mL) of emapalumab after 3 mg/kg dose
  * Cmax values will be calculated using every 48 hour blood collections beginning at the time of emapalumab administration (day 1 after HSCT) until day 21.
Maximum plasma concentration of emapalumab after rescue dosing | Until day 42 or 1 week after rescue dose, whichever is later
  * Measured by the Cmax (ng/mL) of emapalumab after 10mg/kg rescue dose(s).
  * Cmax values will be calculated using every 48 hour blood collections beginning at the time of emapalumab rescue dose administration and continuing for 1 week after the rescue dose.
Number of patients in 10 mg/kg prophylactic dosing arm who maintain CXCL9 levels below the upper limit of normal for the test (</= 647 pg/mL). | Until day 42 or 1 week after rescue dose, whichever is later
  * Measured by plasma CXCL9 levels (pg/mL)
  * CXCL9 levels will be measured every 48 hours beginning at the time of prophylactic emapalumab administration (day 1 after HSCT) and until day 21 after HSCT. Additionally, weekly CXCL9 levels will be obtained from day 21 until day 42 after HSCT.
Number of patients in 3 mg/kg prophylactic dosing arm who maintain CXCL9 levels below the upper limit of normal for the test (</= 647 pg/mL). | Until day 42 or 1 week after rescue dose, whichever is later
  * Measured by plasma CXCL9 levels (pg/mL)
  * CXCL9 levels will be measured every 48 hours beginning at the time of prophylactic emapalumab administration (day 1 after HSCT) and until day 21 after HSCT. Additionally, weekly CXCL9 levels will be obtained from day 21 until day 42 after HSCT.
Number of patients in 10 mg/kg prophylactic dosing arm who maintain CXCL9 levels below 2.6x the upper limit of normal for the test. | Until day 42 or 1 week after rescue dose, whichever is later
  * Measured by plasma CXCL9 levels (pg/mL). This cutoff was chosen based on our prior publication which showed CXCL9 levels above this threshold were associated with graft rejection.
  * CXCL9 levels will be measured every 48 hours beginning at the time of prophylactic emapalumab administration (day 1 after HSCT) and until day 21 after HSCT. Additionally, weekly CXCL9 levels will be obtained from day 21 until day 42 after HSCT.
Number of patients in 3 mg/kg prophylactic dosing arm who maintain CXCL9 levels below 2.6x the upper limit of normal for the test. | Until day 42 or 1 week after rescue dose, whichever is later
  * Measured by plasma CXCL9 levels (pg/mL). This cutoff was chosen based on our prior publication which showed CXCL9 levels above this threshold were associated with graft rejection.
  * CXCL9 levels will be measured every 48 hours beginning at the time of prophylactic emapalumab administration (day 1 after HSCT) and until day 21 after HSCT. Additionally, weekly CXCL9 levels will be obtained from day 21 until day 42 after HSCT.
Emapalumab half-life after 10 mg/kg prophylactic dosing | Until day 42 or time of rescue dose, whichever is sooner
  * Measured using the volume of distribution (L) and clearance (L/h) of emapalumab after 10mg/kg prophylactic dose
  * Half-life will be calculated using every 48 hour sample collections beginning at the time of emapalumab administration (day 1 after HSCT) until day 21. Additionally, weekly blood samples will be obtained from day 21 until day 42 after HSCT.
Emapalumab half-life after 3 mg/kg prophylactic dosing | Until day 42 or time of rescue dose, whichever is sooner
  * Measured using the volume of distribution (L) and clearance (L/h) of emapalumab after 3mg/kg prophylactic dose
  * Half-life will be calculated using every 48 hour sample collections beginning at the time of emapalumab administration (day 1 after HSCT) until day 21. Additionally, weekly blood samples will be obtained from day 21 until day 42 after HSCT.
Emapalumab half-life after 10mg/kg rescue dosing | Until day 42 or time of rescue dose, whichever is sooner
  * Measured using the volume of distribution (L) and clearance (L/h) of emapalumab after 10mg/kg dose(s)
  * Half-life will be calculated using every 48 hour blood collections beginning at the time of emapalumab rescue dose administration and continuing for 1 week after the rescue dose.
Overall survival | 100 days after HSCT.
  • Measured by overall survival of patients who receive prophylactic emapalumab.
Number of patients who develop infections | 100 days after HSCT.
  Measured by the incidence of infection in patients who receive prophylactic emapalumab.
Number of patients who develop mixed chimerism. | 100 days after HSCT.
  Measured by the incidence of mixed chimerism in patients who receive prophylactic emapalumab.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sabulski, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States